CLINICAL TRIAL: NCT03819790
Title: Variability of Glucose Assessed in a Randomized Trial Comparing the Initiation of A Treatment Approach With Biosimilar Basal Insulin Analog Or a Titratable iGlarLixi combinatioN in Type 2 Diabetes Among South Asian Subjects (VARIATION 2 SA Trial)
Brief Title: The Effect of Soliqua on Glucose Variability in Type 2 Patients Among South Asians
Acronym: VARIATION 2 SA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LMC Diabetes & Endocrinology Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VARIATION 2 SA
Record Dates: First submitted 2018-09-24; First posted 2019-01-29 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes, type 2; GLP-1 RA; Insulin glargine; Glucose variability; Insulin Titration; South Asians
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Insulin Glargine; Metformin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into either of two arms by an interactive system in a 1:1 ratio. Randomization will be stratified based on the use of sodium-glucose co-transporter-2 (SGLT2) inhibitors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin Glargine + GLP-1 RA (Experimental): Insulin Soliqua (a titratable combination of insulin Glargine + GLP-1 RA) will be administered at the subject's end-of run-in phase insulin dose (minimum dose of 15 units in both arms) every morning (before first meal of day) and titrate by one unit per day until fasting glucose level of 4-5.5 mmol/L is obtained, with or without metformin.
  Interventions: Drug: Basal insulin glargine and lixisenatide; Drug: Metformin
- Basaglar/Lantus + gliclazide MR (Active Comparator): Basal insulin Basaglar/Lantus will be administered at the subject's end-of run-in phase insulin dose (minimum dose of 15 units in both arms) every morning (before first meal of day) and titrate by one unit per day until fasting glucose level of 4-5.5 mmol/L is obtained, with gliclazide MR 60 mg OD, with or without metformin.
  Interventions: Drug: Basal insulin Basaglar/Lantus + gliclazide MR; Drug: Metformin

INTERVENTIONS:
Drug: Basal insulin glargine and lixisenatide — Soliqua (insulin glargine and lixisenatide): a titratable combination of long-acting basal insulin glargine and lixisenatide (Glucagon-like peptide-1 receptor agonist)
  Arms: Insulin Glargine + GLP-1 RA
Drug: Basal insulin Basaglar/Lantus + gliclazide MR — basal long-acting insulin Basaglar/Lantus with gliclazide MR 60 mg OD
  Arms: Basaglar/Lantus + gliclazide MR
Drug: Metformin — Patients can be administered with most tolerant dose of metformin

SUMMARY:
The overall objective of this study is to compare the effects of Soliqua, a titratable combination of insulin and GLP-1 receptor agonist in a single pen versus Glargine U100 insulin (Basaglar or Lantus) and gliclazide MR, both added to metformin, on measures of glucose variability using masked CGM data among people of South Asian origin living in Canada with type 2 diabetes (T2DM).

DETAILED DESCRIPTION:
The VARIATION 2 SA study is a prospective, open-label, randomized controlled, multi-centre trial to compare the efficacy of two insulin initiation approaches (Soliqua vs Glargine U100 insulin (Basaglar or Lantus) + gliclazide MR) added to maximum tolerated metformin on glucose variability (using masked CGM) in South Asians with T2DM who will initiate insulin therapy with HbA1c of 7.1-11% (inclusive). After giving informed consent and being assessed by eligibility, the patient will stop other oral hypoglycemic agents except metformin (SGLT2 inhibitor may be continued if the patient has cardiovascular diseases history) and enter a 1-week run-in phase with Basaglar or Lantus insulin. During this week (considered as baseline), the patient will: 1) be administered Basaglar or Lantus insulin at an initial dose of 10 units in the morning and increase 1 U/day if fasting glucose >5.5 mmol/L; 2) complete 2 questionnaires to assess the patient-reported outcomes (PROs); 3) wear a masked continuous glucose monitor (CGM) to assess glucose variability; 4) record carbohydrate intake for at least 3 consecutive days. If a patient demonstrates good adherence to Basaglar or Lantus insulin therapy, proper CGM wearing and proper record of carbohydrate intake, and is willing to adhere to insulin treatment will be randomly assigned (1:1) to receive either Soliqua or Glargine U100 insulin (Basaglar or Lantus) + gliclazide MR treatment. The patients will initiate insulin Soliqua or Basaglar/Lantus at their end-of run-in phase insulin dose (minimum dose of 15 units in both arms) every morning (before first meal of day) and titrate by 1 U/day until fasting glucose reaches 4-5.5 mmol/L. In the next 12 weeks, the patients will be optimized their insulin doses via clinic visits or phone calls. They will also be instructed to record their daily fasting glucose, insulin dose, hypoglycemic episodes and any adverse events in a logbook. The primary outcome is to compare the difference of average percentage of Time in Range (4.0-10.0 mmol/L) within 24 hours over the CGM period between two treatments at week 13 after randomization. The co-primary is to compare the difference average percentage of Time in Range (4.0-10.0 mmol/L) within 12 hours (6 AM- 6 PM) over the CGM period between two treatments at week 13 after randomization. The secondary outcomes include the differences on other measurements of glucose variability and patient-reported outcomes (PROs).

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults with clinical diagnosis of T2DM diagnosed at least 1 year before screening and in stable health as assessed by investigator
* Age between 18 and 80 years (inclusive)
* Body mass index (BMI) between 20-40 kg/m2 (inclusive)
* South Asian origin including Afghanistani, Bangladeshi, Indian, Nepali, Pakistani and Sri Lankan. This includes those patients who identify themselves as South Asian origin because their ancestors moved from South Asian to another country (e.g. Caribbean islands, Fiji, etc.)
* A1C in range of 7.1-11% (inclusive)
* Fasting glucose on self-monitoring of blood glucose (SMBG) or laboratory testing < 15 mmol/L within the last 30 days
* Insulin naïve, uncontrolled on oral hypoglycemic medications
* Kidney function assessment with eGFR >30 mL/min/1.73 m2
* Written informed consent obtained

Exclusion Criteria:

* History of insulin use (except emergency short-term use defined as less than 12 weeks for acute illness, hospitalization, pregnancy or with steroid use)
* Use of GLP-1 receptor agonist in the past 3 months
* Previous discontinuation of a GLP-1 receptor agonist due to safety, tolerability or lack of efficacy
* Pregnant or anticipating pregnancy
* Current use of steroid
* Currently on any supervised, intensive, weight-loss dietary or exercise program
* History of gastroparesis with moderate or higher severity
* History of pancreatitis
* Amylase and /or lipase more than three times the upper limit of normal or calcitonin ≥ 20 pg/mL (5.9 pmol/L)
* Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia (MEN) syndrome
* Allergic reaction to insulin secretagogues
* History of weight loss surgery (bariatric bypass surgery or gastric banding)
* Inability to check SMBG or wear CGM
* History of severe liver disease or alcohol abuse
* Severe hypoglycemic reaction (defined as third-party or ambulance assistance or emergency department visit) within the last 3 months before screening visit
* Night-shift workers
* Patients who are recommended to achieve relaxed targets of A1C up to 8.5% by Diabetes Canada 2018 clinical practice guidelines
* Current enrollment in another intervention study
* Patients who miss ≥1 injections of Basaglar/Lantus or discontinue the CGM device or can not record carbohydrate intake correctly during the run-in phase

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Time in range at week 13 | 7 days
  Time with CGM glucose between 4.0 - 10.0 mmol/L within 24 hours over the 7-day CGM period at week 13 after randomization
Time in range within 12-hours (6 AM -6 PM) at week 13 | 7 days
  Time with CGM glucose between 4.0 - 10.0 mmol/L within 12-hours (6 AM -6 PM) over the 7-day CGM period at week 13 after randomization

SECONDARY OUTCOMES:
Daily glucose standard deviation (SD) at week 13 | 7 days
  Daily SD of CGM glucose over the 7-day CGM period at week 13 after randomization
Overall SD of CGM glucose at week 13 | 7 days
  Overall SD of CGM glucose over the 7-day CGM period at week 13 after randomization
Mean of glucose at week 13 | 7 days
  Mean of CGM glucose over the 7-day CGM period at week 13 after randomization
Frequency of hypoglycemia at week 13 | 7 days
  Number of hypoglycemic event which is defined as CGM glucose <4.0 mmol/L for at least 15 mins (3 consecutive CGM readings) over the 7-day CGM period at week 13 after randomization
Time in hypoglycemia at week 13 | 7 days
  Time with CGM glucose < 4.0 mmol/L over the 7-day CGM period at week 13 after randomization
Frequency of hyperglycemia at week 13 | 7 days
  Number of hyperglycemic event which is defined as CGM glucose >10.0 mmol/L at least 15 mins (3 consecutive CGM readings) over the 7-day CGM period at week 13 after randomization
Time in hyperglycemia at week 13 | 7 days
  Time with CGM glucose >10.0 mmol/L over the 7-day CGM period at week 13 after randomization
Daily glucose standard deviation (SD) within 12 hours (6AM-6PM) at week 13 | 7 days
  Daily SD of CGM glucose within 12 hours (6AM-6PM) over the 7-day CGM period at week 13 after randomization
Overall SD of glucose within 12 hours (6AM-6PM) at week 13 | 7 days
  Overall SD of CGM glucose within 12 hours (6AM-6PM) over the 7-day CGM period at week 13 after randomization
Mean of glucose within 12 hours (6AM-6PM) at week 13 | 7 days
  Mean of CGM glucose within 12 hours (6AM-6PM) over the 7-day CGM period at week 13 after randomization
Frequency of hypoglycemia within 12 hours (6AM-6PM) at week 13 | 7 days
  Number of hypoglycemic event which is defined as CGM glucose <4.0 mmol/L for at least 15 mins (3 consecutive CGM readings) within 12 hours (6AM-6PM) over the 7-day CGM period at week 13 after randomization
Time in hypoglycemia within 12 hours (6AM-6PM) at week 13 | 7 days
  Time with CGM glucose <4.0 mmol/L within 12 hours (6AM-6PM) over the 7-day CGM period at week 13 after randomization
Frequency of hyperglycemia within 12 hours (6AM-6PM) at week 13 | 7 days
  Number of hypoglycemic event which is defined as CGM glucose >10.0 mmol/L for at least 15 mins (3 consecutive CGM readings) within 12 hours (6AM-6PM) over the 7-day CGM period at week 13 after randomization
Time in hyperglycemia within 12 hours (6AM-6PM) at week 13 | 7 days
  Time with CGM glucose >10.0 mmol/L within 12 hours (6AM-6PM) over the 7-day CGM period at week 13 after randomization
A1C mean at week 13 | Week 13
  Average of A1C at week 13 after randomization
Changes A1C | 15 weeks
  A1C value at Visit10 at 13 weeks after randomization minus A1C value at Visit 1 at week -2 (2 weeks before randomization)
Proportion of A1C <7% at week 13 | Week 13
  the number of patients who have A1C <7% divided by the total number of patients who have A1C measurement at week 13 after randomization
Proportion of A1C <8% at week 13 | Week 13
  the number of patients who have A1C <8% divided by the total number of patients who have A1C measurement at week 13 after randomization
Mean basal insulin dose at week 13 | Week 13
  Average of basal insulin dose from patients' diary at week 13 after randomization
Change in weight | 15 weeks
  Weight difference between week 13 after randomization and baseline at week -2 (2 weeks before randomization) = weight at Visit 10 at week 13 - weight at Visit 1 at week -2.
Change in waist circumference | 15 weeks
  Waist circumference change between week 13 after randomization and baseline at week -2 (2 week before randomization)= waist circumference at Visit 10 at week 13- waist circumference at Visit 1 at week -2
Change in carbohydrate intake | 14 weeks
  Carbohydrate intake change between week 13 after randomization and baseline at week -1 = carbohydrate intake at Visit 10 at week 13 - carbohydrate intake at Visit 2 at week -1 (1 week before randomization)
Proportion of patients who have A1C ≤ 7% with no hypoglycemia and no weight gain from baseline | Week 13
  the number of patients who have A1C ≤ 7% with no hypoglycemia and no weight gain from baseline divided by the total number of patients at Week 13 after randomization
Proportion of patients who have A1C ≤ 7% with no hypoglycemia and weight gain <3% from baseline | Week 13
  the number of patients who have A1C ≤ 7% with no hypoglycemia and weight gain <3% from baseline divided by the total number of patients at Week 13 after randomization
Proportion of patients who have fasting blood glucose ≤ 5.5 mmol/L without nocturnal hypoglycemia | Week 13
  the number of patients who have fasting blood glucose ≤ 5.5 mmol/L without nocturnal hypoglycemia divided by the total number of patients at Week 13 after randomization
Change in DiabMedSat Score | 14 weeks
  DiabMedSat Score will be generated using Diabetes Medication Satisfaction (DiabMedSat) questionnaire. It measures the levels of the subjects' satisfaction with their diabetes medication(s). The range of the score is 0 to 100. The higher the score, the greater the satisfaction. The changes in the score will measure the score difference between Visit 10 at week 13 after randomization and Visit 2 at week -1 (1 week before randomization)
Change in HFS Score | 14 weeks
  HFS Score will be measured by the Hypoglycemia Fear Survey which assesses the subject's behaviors to avoid hypoglycemia and to measure the subjects' worries about hypoglycemia and its consequences in the past 3 months. The range of the score will be 0 to 132. The higher the score, the greater the fear.
  The changes will be the score difference between Visit 10 at week 13 after randomization and Visit 2 at week -1 (1 week before randomization).
HCP treatment satisfaction score | Week 13
  HCP treatment satisfaction score will be generated from Healthcare Provider treatment satisfaction questionnaire. It measures the levels of satisfaction of physicians in this study when prescribing this medication at Visit 10 at week 13 after randomization. The range is 0 to 15. The higher the score, the greater the satisfaction.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - LMC Brampton, Brampton, Ontario
  - LMC Etobicoke, Etobicoke, Ontario
  - LMC Scarborough, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Lipska KJ, Yao X, Herrin J, McCoy RG, Ross JS, Steinman MA, Inzucchi SE, Gill TM, Krumholz HM, Shah ND. Trends in Drug Utilization, Glycemic Control, and Rates of Severe Hypoglycemia, 2006-2013. Diabetes Care. 2017 Apr;40(4):468-475. doi: 10.2337/dc16-0985. Epub 2016 Sep 22. PMID 27659408
- [Background] Tobias DK, Pan A, Jackson CL, O'Reilly EJ, Ding EL, Willett WC, Manson JE, Hu FB. Body-mass index and mortality among adults with incident type 2 diabetes. N Engl J Med. 2014 Jan 16;370(3):233-44. doi: 10.1056/NEJMoa1304501. PMID 24428469
- [Background] Scheen AJ, Van Gaal LF. Combating the dual burden: therapeutic targeting of common pathways in obesity and type 2 diabetes. Lancet Diabetes Endocrinol. 2014 Nov;2(11):911-22. doi: 10.1016/S2213-8587(14)70004-X. Epub 2014 Feb 19. PMID 24731666
- [Background] Degn KB, Brock B, Juhl CB, Djurhuus CB, Grubert J, Kim D, Han J, Taylor K, Fineman M, Schmitz O. Effect of intravenous infusion of exenatide (synthetic exendin-4) on glucose-dependent insulin secretion and counterregulation during hypoglycemia. Diabetes. 2004 Sep;53(9):2397-403. doi: 10.2337/diabetes.53.9.2397. PMID 15331551
- [Background] Degn KB, Juhl CB, Sturis J, Jakobsen G, Brock B, Chandramouli V, Rungby J, Landau BR, Schmitz O. One week's treatment with the long-acting glucagon-like peptide 1 derivative liraglutide (NN2211) markedly improves 24-h glycemia and alpha- and beta-cell function and reduces endogenous glucose release in patients with type 2 diabetes. Diabetes. 2004 May;53(5):1187-94. doi: 10.2337/diabetes.53.5.1187. PMID 15111485
- [Background] Flint A, Raben A, Astrup A, Holst JJ. Glucagon-like peptide 1 promotes satiety and suppresses energy intake in humans. J Clin Invest. 1998 Feb 1;101(3):515-20. doi: 10.1172/JCI990. PMID 9449682
- [Background] Leiter LA, Nauck MA. Efficacy and Safety of GLP-1 Receptor Agonists Across the Spectrum of Type 2 Diabetes Mellitus. Exp Clin Endocrinol Diabetes. 2017 Jul;125(7):419-435. doi: 10.1055/s-0043-103969. Epub 2017 Jul 19. German. PMID 28724168
- [Background] Zaccardi F, Htike ZZ, Webb DR, Khunti K, Davies MJ. Benefits and Harms of Once-Weekly Glucagon-like Peptide-1 Receptor Agonist Treatments: A Systematic Review and Network Meta-analysis. Ann Intern Med. 2016 Jan 19;164(2):102-13. doi: 10.7326/M15-1432. Epub 2015 Dec 8. PMID 26642233
- [Background] Rosenstock J, Fonseca VA, Gross JL, Ratner RE, Ahren B, Chow FC, Yang F, Miller D, Johnson SL, Stewart MW, Leiter LA; Harmony 6 Study Group. Advancing basal insulin replacement in type 2 diabetes inadequately controlled with insulin glargine plus oral agents: a comparison of adding albiglutide, a weekly GLP-1 receptor agonist, versus thrice-daily prandial insulin lispro. Diabetes Care. 2014 Aug;37(8):2317-25. doi: 10.2337/dc14-0001. Epub 2014 Jun 4. PMID 24898300
- [Background] Diamant M, Nauck MA, Shaginian R, Malone JK, Cleall S, Reaney M, de Vries D, Hoogwerf BJ, MacConell L, Wolffenbuttel BH; 4B Study Group. Glucagon-like peptide 1 receptor agonist or bolus insulin with optimized basal insulin in type 2 diabetes. Diabetes Care. 2014 Oct;37(10):2763-73. doi: 10.2337/dc14-0876. Epub 2014 Jul 10. PMID 25011946
- [Background] Writing Group for the DCCT/EDIC Research Group; Orchard TJ, Nathan DM, Zinman B, Cleary P, Brillon D, Backlund JY, Lachin JM. Association between 7 years of intensive treatment of type 1 diabetes and long-term mortality. JAMA. 2015 Jan 6;313(1):45-53. doi: 10.1001/jama.2014.16107. PMID 25562265
- [Background] Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008 Oct 9;359(15):1577-89. doi: 10.1056/NEJMoa0806470. Epub 2008 Sep 10. PMID 18784090
- [Background] Lind M, Svensson AM, Kosiborod M, Gudbjornsdottir S, Pivodic A, Wedel H, Dahlqvist S, Clements M, Rosengren A. Glycemic control and excess mortality in type 1 diabetes. N Engl J Med. 2014 Nov 20;371(21):1972-82. doi: 10.1056/NEJMoa1408214. PMID 25409370
- [Background] Esposito K, Giugliano D, Nappo F, Marfella R; Campanian Postprandial Hyperglycemia Study Group. Regression of carotid atherosclerosis by control of postprandial hyperglycemia in type 2 diabetes mellitus. Circulation. 2004 Jul 13;110(2):214-9. doi: 10.1161/01.CIR.0000134501.57864.66. Epub 2004 Jun 14. PMID 15197140
- [Background] Kilpatrick ES, Rigby AS, Atkin SL. A1C variability and the risk of microvascular complications in type 1 diabetes: data from the Diabetes Control and Complications Trial. Diabetes Care. 2008 Nov;31(11):2198-202. doi: 10.2337/dc08-0864. Epub 2008 Jul 23. PMID 18650371
- [Background] Bajaj HS, Venn K, Ye C, Patrick A, Kalra S, Khandwala H, Aslam N, Twum-Barima D, Aronson R. Lowest Glucose Variability and Hypoglycemia Are Observed With the Combination of a GLP-1 Receptor Agonist and Basal Insulin (VARIATION Study). Diabetes Care. 2017 Feb;40(2):194-200. doi: 10.2337/dc16-1582. Epub 2016 Dec 2. PMID 27913575
- [Background] Chiu M, Austin PC, Manuel DG, Tu JV. Comparison of cardiovascular risk profiles among ethnic groups using population health surveys between 1996 and 2007. CMAJ. 2010 May 18;182(8):E301-10. doi: 10.1503/cmaj.091676. Epub 2010 Apr 19. PMID 20403888
- [Background] Chiu M, Maclagan LC, Tu JV, Shah BR. Temporal trends in cardiovascular disease risk factors among white, South Asian, Chinese and black groups in Ontario, Canada, 2001 to 2012: a population-based study. BMJ Open. 2015 Aug 10;5(8):e007232. doi: 10.1136/bmjopen-2014-007232. PMID 26260346
- [Background] Gujral UP, Pradeepa R, Weber MB, Narayan KM, Mohan V. Type 2 diabetes in South Asians: similarities and differences with white Caucasian and other populations. Ann N Y Acad Sci. 2013 Apr;1281(1):51-63. doi: 10.1111/j.1749-6632.2012.06838.x. Epub 2013 Jan 14. PMID 23317344
- [Background] Yale JF, Berard L, Groleau M, Javadi P, Stewart J, Harris SB. TITRATION: A Randomized Study to Assess 2 Treatment Algorithms with New Insulin Glargine 300 units/mL. Can J Diabetes. 2017 Oct;41(5):478-484. doi: 10.1016/j.jcjd.2017.06.007. Epub 2017 Aug 10. PMID 28803820
- [Derived] Bajaj HS, Chu L, Bansal N, Brown RE, Dhillon G, Gupta R, Bhela JS, Padda JK, Khandwala H, Venn K, Aronson R. Randomized Comparison of Initiating the Fixed-Ratio Combination of iGlarLixi or Biosimilar Insulin Glargine Together With Gliclazide in Participants of South Asian Origin With Type 2 Diabetes: VARIATION 2 SA Trial. Can J Diabetes. 2022 Jul;46(5):495-502. doi: 10.1016/j.jcjd.2022.02.003. Epub 2022 Feb 11. PMID 35752566